CLINICAL TRIAL: NCT06102109
Title: Long-term Results of Two Surgical Methods for Scleral IOL Implantation and Fixation in Eyes Without Capsular Support: Yamane- Versus 4-flanged Technique
Acronym: YAMPOINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Claudette Abela-Formanek, Univ. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y4P0923
Record Dates: First submitted 2023-09-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Lens Luxation; IOL Subluxation; IOL Opacification; Aphakia - No Lens Capsule
Keywords: Scleral fixated IOL; Yamane; 4 flanged technique
MeSH Terms: conditions — Lens Subluxation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yamane Arm (Active Comparator): Scleral IOL fixation using the Yamane technique. A 3 piece IOL (Kowa Avansee Preset) gets fixated in the sclera.
  Interventions: Procedure: Pars plana vitrectomy; Procedure: IOL explantation; Procedure: Scleral IOL fixation Yamane Technique
- "4-flanged" Arm (Active Comparator): Scleral IOL fixation using the 4 flanged technique. A 4 loop haptic IOL (Physiol Micropure 123) gets fixated in the sclera using 6.0 polypropylene suture
  Interventions: Procedure: Pars plana vitrectomy; Procedure: IOL explantation; Procedure: Scleral IOL fixation "4-flanged" Technique

INTERVENTIONS:
Procedure: Pars plana vitrectomy — 25gauge pars plana vitrectomy: to remove the vitreous if present
Procedure: IOL explantation — Removing if present a subluxated IOL from the anterior chamber or the vitreous cavity
Procedure: Scleral IOL fixation Yamane Technique — Scleral IOL fixation using the Yamane technique. A 3 piece IOL (Kowa Avansee Preset) gets fixated in the sclera using only its haptics, which are externalised 2.5mm behind the blue line. The haptic ends are flanged using a thermo cautery to prevent slipping back in.
  Arms: Yamane Arm
Procedure: Scleral IOL fixation "4-flanged" Technique — Scleral IOL fixation using the 4 flanged technique. A 4 loop haptic IOL (Physical Micropure 123) gets fixated in the sclera using one 6.0 polypropylene suture per 2 haptic loops, which are put trough the loops in a W shape. The suture ends are externalised 2.5mm behind the blue line and its ends are flanged using a thermo cautery to prevent slipping back in.
  Arms: "4-flanged" Arm

SUMMARY:
This study is a comparison of the surgical techniques and postoperative outcome between the two intrascleral IOL fixation techniques: Yamane technique versus the 4-flanged technique.

The main objectives are postoperative lens tilt, duration of surgery, intra- and postoperative complication rates and scleral integrity around the flanges.

ELIGIBILITY:
Inclusion Criteria:

* - Necessity for IOL (re)fixation in the absence of capsular support
* willing to give informed consent and follow-up the duration of study

Exclusion Criteria:

* Anatomical or other contraindications for suture less IOL fixation, such as presence of a trabeculectomy bleb or scleromalacia
* active inflammatory diseases of the eye

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
IOL tilt | 3 years
  The postoperative intra ocular lens tilt in degree measured by an anterior segment optical coherence tomography device (Casia 2, Tommy, Japan)
IOL decentration | 3 years
  The postoperative intra ocular lens decentration in millimetres measured by an anterior segment optical coherence tomography device (Casia 2, Tommy, Japan)

SECONDARY OUTCOMES:
Best corrected visual outcome | 12 weeks
  The achieved best corrected visual (in Snellen) outcome after Intraocular lens implantation
Flange erosion and intrusion | 3 years
  Risks of flange erosion trough the conjuctiva or intrusion through the sclera over the investigated time period

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided